CLINICAL TRIAL: NCT02510313
Title: Effectiveness Trial of a Family Home Visiting Intervention to Promote Early Child Development Among Families Served by the Social Protection System in Rwanda
Brief Title: Strong Families, Thriving Children "Sugira Muryango"_Activity C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Responsible Party: Principal Investigator, Theresa Betancourt, Salem Professor in Global Practice, Boston College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB16-1570
Record Dates: First submitted 2015-07-26; First posted 2015-07-29 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Child Development, Social Protection

STUDY DESIGN:
Intervention Model Description: The proposed study design consists of a four-arm cluster randomized control trial (CRT), which will span approximately 52 cells in 3 districts of Rwanda to compare outcomes among VUP eligible households with at least one child 6-36 months in the following study arms:
  * Classic VUP public works (control)
  * Expanded VUP public works (control)
  * Combined Classic VUP public works with Sugira Muryango (treatment)
  * Combined Expanded VUP public works with Sugira Muryango (treatment)
Who Masked: Outcomes Assessor
Masking Description: Our study works with Laterite to oversee data collection in the field. Laterite enumerators are blind to study condition and therefore do not know which study arm, apart from their VUP status (class or expanded), participants have been randomized into.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Classic VUP (Control) (No Intervention): Families receive benefits (cash) in exchange for state-sanctioned labour intensive work.
- Expanded VUP (No Intervention): Families receive benefits (cash) in exchange for state-sanctioned flexible labour within close proximity (2 km) to household. Eligible for variation of minimum graduation package benefits, such as asset transfer, financial literacy, skills training, sensitizations.
- Sugira Muryango & Classic VUP (Experimental): Families receive combination of Sugira Muryango and benefits (cash) in exchange for state-sanctioned labour intensive work.
  Interventions: Other: Sugira Muryango
- Sugira Muryango & Expanded VUP (Experimental): Families receive combination of Sugira Muryango and benefits (cash) in exchange for state-sanctioned flexible labour within close proximity (2 km) to household. Eligible for variation of minimum graduation package benefits, such as asset transfer, financial literacy, skills training, sensitizations.
  Interventions: Other: Sugira Muryango

INTERVENTIONS:
Other: Sugira Muryango — Strong Families, Thriving Children "Sugira Muryango" is a home-visiting intervention that empowers low-income families enrolled in Rwanda's social protection system to support early childhood development and healthy family functioning.
  Arms: Sugira Muryango & Classic VUP; Sugira Muryango & Expanded VUP

SUMMARY:
The proposed study will test the effectiveness of the Strong Families, Thriving Children "Sugira Muryango" program as delivered by community based workers and aligned with the Rwandan social protection system. Sugira Muryango is a preventive, family-based model that uses home visiting and coaching to encourage responsive parent-child interactions and discourage violence and harsh punishment targeting families living in extreme poverty. Integration of scalable, cost-effective interventions into poverty-reduction and other social welfare programs has great potential as an effective means to promote child development and reduce familial violence and in a range of culturally diverse, low-resource settings.

DETAILED DESCRIPTION:
Globally, more than 200 million children may not reach their full developmental potential due to poverty and adversity. This is most evident in World Bank-classified Low- and Middle-Income Countries (LMICs) struggling with the confluence of war, community violence, poverty and disease. Research across a range of cultures and settings finds that children living in compounded adversity face increased risks of poor child development outcomes and emotional and behavioral problems that can perpetuate a cycle of poverty and violence. Integrated programs and family-based interventions for promoting child development, healthy parent-child relationships and reducing household violence affecting children are insufficiently tested in culturally diverse and low-resource settings despite compelling data about such risks. The proposed study will investigate the effectiveness of the Sugira Muryango program as an innovative approach to early childhood development promotion. Sugira Muryango is a preventive, family-based model that uses home visiting and caregiver coaching; it encourages responsive caregiver-child interactions and discourages violence and harsh punishment among families living in extreme poverty. By providing home-based coaching that helps parents manage stress, reduce harsh punishment and engage in responsive parenting with early childhood stimulation, it is possible to effect improvements in parent-child relationships and child development outcomes. Sugira Muryango will be implemented alongside Rwanda's flagship poverty reduction initiative, Vision 2020 Umurenge Program (VUP). Classic VUP components mainly focus on cash-for-work on labor intensive public works projects. With government and development partner support, VUP is piloting a more enhanced public works model that has child and gender sensitive components, with flexible public works options that are closer to beneficiary households. Along such the expanded public works program currently under pilot by VUP, a minimum graduation package is also available, which is providing additional variables of financial literacy, asset transfers, skills training, and sensitizations surrounding a range of topics (e.g., education, health, nutrition).

A four-arm cluster randomized trial (CRT) will enroll 1,040 VUP-eligible families with children aged 6-36 months to compare outcomes among children and parents in families receiving: (1) Control/Classic VUP, (2) Expanded VUP, (3) Combined Classic VUP plus Sugira Muryango and (4) Combined Expanded VUP plus Sugira Muryango. A cost analysis will provide practical information on the feasibility and cost of integrating Sugira Muryango into VUP programming and a process evaluation will produce useful implementation tools for dissemination and scale-up.

Study Aims are to (1) assess effectiveness of Sugira Muryango in promoting responsive parenting, reducing violence and harsh punishment and promoting early child development in families living in poverty; (2) to assess the interaction between Sugira Muryano and classic/expanded VUP programming and (3) to assess costs, barriers and facilitators of integrating the Sugira Muryango package into VUP or other government programming, such as the Ministry of Gender and Family Promotion (MIGEPROF), which holds the early childhood development mandate. This initiative seeks to promote cross sectoral and ministerial collaboration, a key pillar of the Government of Rwanda.

ELIGIBILITY:
Beneficiary Inclusion Criteria:

- All participants must live in chosen District(s) of Rwanda.

Inclusion criteria for families are:

1. being VUP-eligible
2. having at least one children aged 0-6 years living in the home
3. having caregiver willing to discuss and enhance their parenting practices by interacting with a home-visiting coach.

Caregiver eligibility:

1. is aged 18 or older and cares for child(ren)
2. lives in the same household as child(ren). We will enroll both single and dual caregiver families to reflect population dynamics. Legal guardians may be aunts, uncles, grandparents, or foster parents.

Exclusion Criteria:

* do not live in chosen District of Rwanda
* do not have children between the ages of 0 and 6 years living in their household for whom they are the primary caregiver
* they are not enrolled in Rwanda's public works social protection program VUP, or have severe cognitive impairments which preclude their ability to speak to the research questions under study
* families in the midst of crisis (e.g., a caregiver with active suicidal attempts or psychosis) and refer them to appropriate services.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2911 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in parent-child relationship | Years 2 & 3
  Questionnaires and observations will be used to assess this outcome
Change from baseline in responsive caregiving practices | Years 2 & 3
  Questionnaires and observations will be used to assess this outcome
Change from baseline in child development | Years 2 & 3
  Questionnaires and observations will be used to assess this outcome
Change from baseline in violence in the home | Years 2 & 3
  Questionnaires will be used to assess this outcome
Change from baseline in child health and nutrition | Years 2 & 3
  Questionnaires and observations will be used to assess this outcome

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Betancourt, Sc.D, Principal Investigator — Boston College School of Social Work
Locations (1):
- FXB Rwanda, Kigali, Rwanda

REFERENCES:
- [Background] Shonkoff JP. Building a new biodevelopmental framework to guide the future of early childhood policy. Child Dev. 2010 Jan-Feb;81(1):357-67. doi: 10.1111/j.1467-8624.2009.01399.x. PMID 20331672
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Dyregrov A, Gupta L, Gjestad R, Mukanoheli E. Trauma exposure and psychological reactions to genocide among Rwandan children. J Trauma Stress. 2000 Jan;13(1):3-21. doi: 10.1023/A:1007759112499. PMID 10761171
- [Background] Betancourt TS, Ng LC, Kirk CM, Munyanah M, Mushashi C, Ingabire C, Teta S, Beardslee WR, Brennan RT, Zahn I, Stulac S, Cyamatare FR, Sezibera V. Family-based prevention of mental health problems in children affected by HIV and AIDS: an open trial. AIDS. 2014 Jul;28 Suppl 3(0 3):S359-68. doi: 10.1097/QAD.0000000000000336. PMID 24991909
- [Derived] Jensen SGK, Placencio-Castro M, Murray SM, Littman J, Bazubagira SM, Uwizeye D, Sezibera V, Betancourt TS. Four-year follow-up to a home-visiting intervention to promote early childhood development and prevent family violence in rural Rwanda: the Sugira Muryango cluster randomised trial. BMJ Glob Health. 2025 Jun 8;10(6):e017866. doi: 10.1136/bmjgh-2024-017866. PMID 40484411
- [Derived] Jensen SK, Placencio-Castro M, Murray SM, Brennan RT, Goshev S, Farrar J, Yousafzai A, Rawlings LB, Wilson B, Habyarimana E, Sezibera V, Betancourt TS. Effect of a home-visiting parenting program to promote early childhood development and prevent violence: a cluster-randomized trial in Rwanda. BMJ Glob Health. 2021 Jan;6(1):e003508. doi: 10.1136/bmjgh-2020-003508. PMID 33514591
- [Derived] Betancourt TS, Jensen SKG, Barnhart DA, Brennan RT, Murray SM, Yousafzai AK, Farrar J, Godfroid K, Bazubagira SM, Rawlings LB, Wilson B, Sezibera V, Kamurase A. Promoting parent-child relationships and preventing violence via home-visiting: a pre-post cluster randomised trial among Rwandan families linked to social protection programmes. BMC Public Health. 2020 May 6;20(1):621. doi: 10.1186/s12889-020-08693-7. PMID 32375840

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT02510313/Prot_SAP_000.pdf